CLINICAL TRIAL: NCT00580112
Title: Phase II, Multicenter, Open-label, Clinical Trial of Trabectedin (Yondelis) in Metastatic Breast Cancer Patients With Triple Negative Profile (ER-, PR-, HER2-), HER2 Overexpressing Tumors and BRCA1 or BRCA2 Mutation Carriers
Brief Title: An Efficacy Study of Trabectedin in the Treatment of Participants With Specific Subtypes of Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014764; ET-B-027-06 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Breast Neoplasms
Keywords: Breast Neoplasms; Trabectedin; Yondelis
MeSH Terms: conditions — Breast Neoplasms | interventions — Dexamethasone; Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): Participants with triple negative phenotype: estrogen receptor, progesterone receptor and human estrogen receptor-2 (HER-2) negative status for breast cancer (abnormal tissue that grows and spreads in the body until it kills) will receive trabectedin 1.3 milligram per meter square (mg/m^2) intravenous infusion (a fluid or a medicine delivered into a vein by way of a needle) over 3-hours (hrs) every 3 weeks, on Day 1 of each cycle. Each cycle length will be 3 weeks. Treatment will be continued until disease progression, unmanageable toxicity, participant refusal or treatment delay no longer than 3 weeks due to toxicity. Along with study drug participants will be given dexamethasone 4 milligram (mg) orally 24 hrs and 12hrs before study drug infusion on Day -1, followed by dexamethasone 20 mg intravenously 30 minutes before study drug infusion on Day 1, followed by dexamethasone 4 mg orally 24, 36, 48, 60 and 72hrs after the start of study drug infusion from Day 1 to 3.
  Interventions: Drug: Dexamethasone; Drug: Trabectedin
- Group B (Experimental): Participants with overexpressing HER-2 breast cancer will receive trabectedin 1.3 mg/m^2 intravenous infusion over 3-hrs every 3 weeks, on Day 1 of each cycle. Each cycle length will be 3 weeks. Treatment will be continued until disease progression, unmanageable toxicity, participant refusal or treatment delay no longer than 3 weeks due to toxicity. Along with study drug participants will be given dexamethasone 4 milligram (mg) orally 24 hrs and 12hrs before study drug infusion on Day -1, followed by dexamethasone 20 mg intravenously 30 minutes before study drug infusion on Day 1, followed by dexamethasone 4 mg orally 24, 36, 48, 60 and 72 hrs after the start of study drug infusion from Day 1 to 3.
  Interventions: Drug: Dexamethasone; Drug: Trabectedin
- Group C (Experimental): Participants with familial breast cancer gene 1 (BRCA1) or breast cancer gene 2 (BRCA2) mutation carriers cancer will receive trabectedin 1.3 mg/m^2 intravenous infusion over 3-hrs every 3 weeks on Day 1 of each cycle. Each cycle length will be 3 weeks. Treatment will be continued until disease progression, unmanageable toxicity, participant refusal or treatment delay no longer than 3 weeks due to toxicity. Along with study drug participants will be given dexamethasone 4 mg orally 24 hrs and 12hrs before study drug infusion on Day -1, followed by dexamethasone 20 mg intravenously 30 minutes before study drug infusion on Day 1, followed by dexamethasone 4 mg orally 24, 36, 48, 60 and 72 hrs after the start of study drug infusion from Day 1 to 3.
  Interventions: Drug: Dexamethasone; Drug: Trabectedin

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 4 mg orally 24 hrs and 12 hrs before study drug infusion on Day -1, followed by dexamethasone 20 mg intravenously 30 minutes before study drug infusion on Day 1, followed by dexamethasone 4 mg orally 24, 36, 48, 60 and 72 hrs after the start of study drug infusion on Day 1 to 3.
Drug: Trabectedin — Trabectedin 1.3 mg/m^2 intravenous infusion over 3-hrs every 3 weeks, on Day 1 of each cycle. Each cycle length will be 3 weeks.
  Other Names: Yondelis

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of trabectedin in 3 subpopulations of participants with previously treated progressive metastatic ( spread of a cancer from one organ or part to another non-adjacent organ or part) breast cancer (abnormal tissue that grows and spreads in the body until it kills) participants.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), prospective (study following participants forward in time), multi-center (when more than 1 hospital or medical school team work on a medical research study) study evaluating the effectiveness and safety of trabectedin in 3 subpopulations of breast cancer participants: Group A: triple negative profile for estrogen receptor, progesterone receptor and human estrogen receptor, Group B: human epidermal growth factor receptor-2 overexpressing tumors (HER-2+) and Group C: familial breast cancer gene 1 (BRCA1) or breast cancer gene 2 (BRCA2) mutation carrier. Participants will receive trabectedin 1.3 milligram per square meter (mg/m^2) intravenous infusion (a fluid or a medicine delivered into a vein by way of a needle) over 3-hour every 3 weeks, on Day 1 of each cycle. Each cycle length will be 3 weeks. Treatment will be continued until disease progression, unmanageable toxicity, participant refusal or treatment delay no longer than 3 weeks due to toxicity. Efficacy will be primarily evaluated by percentage of participants with confirmed objective response by independent external review and Investigators assessment. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically proven diagnosis of progressive metastatic breast cancer
* Participants with measurable disease as per the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines
* Participants with bone metastases currently receiving bisphosphonates for palliation will be eligible if other sites of measurable disease are present
* Participants with Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1 and adequately recovered from the acute toxicity of any prior treatment
* Participants with serum creatinine less than or equal to 1.5 milligram per deciliter (mg/dl) or creatinine clearance greater than or equal to 30 milliliter per minute (ml/min)

Exclusion Criteria:

* Participants with previous exposure to trabectedin
* Participants with more than 3 previous chemotherapy regimens for metastatic disease and known hypersensitivity to components of trabectedin intravenous formulation or dexamethasone
* Pregnant or lactating women or any women of childbearing potential who is not employing adequate contraception
* Completion of previous therapy : Less than 2 weeks from radiation therapy or last dose of hormonal therapy, less than 3 weeks from previous biological therapy or chemotherapy
* Participants with known leptomeningeal disease and other serious illnesses like congestive heart failure or angina pectoris; myocardial infarction within 1 year before enrolment; uncontrolled arterial hypertension or arrhythmias or active infection or psychiatric disorder or active viral hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2007-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Confirmed Objective Response (OR) by Independent External Review (IER) | Baseline up to progressive disease or death, assessed every 6 weeks (up to 90 weeks)
  Percentage of participants with confirmed objective response will be based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR is defined as disappearance of all target lesions. PR is those with at least 30 percent decrease in the sum of longest dimensions of target lesions taking as a reference baseline sum longest dimensions. IER will be done to re-examine all Investigator assessed outcomes.
Percentage of Participants With Confirmed Objective Response (OR) by Investigators' Assessment | Baseline up to progressive disease or death, assessed every 6 weeks (up to 90 weeks)
  Percentage of participants with objective response based assessment of confirmed CR or confirmed PR according to RECIST. Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. The CR is defined as disappearance of all target lesions. The PR is those with at least 30 percent decrease in the sum of longest dimensions of target lesions taking as a reference baseline sum longest dimensions.

SECONDARY OUTCOMES:
Duration of Response (DR) by Independent Expert Review (IER) | Baseline up to progressive disease or death, assessed every 6 weeks (up to 90 weeks)
  Duration of Response is considered as time in months from the first documentation of objective tumor response to objective tumor progression or death due to any cause. Duration of tumor response was calculated as: (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that will be subsequently confirmed plus 1) divided by 30.44. DR will be calculated for the subgroup of participants with a confirmed objective tumor response. IER will be done to re-examine all Investigator assessed outcomes and to provide an independent assessment of response and progression date.
Duration of Response (DR) by Investigators' Assessment | Baseline up to progressive disease or death, assessed every 6 weeks (up to 90 weeks)
  Duration of Response is considered as time in months from the first documentation of objective tumor response to objective tumor progression or death due to any cause. Duration of tumor response is calculated as: (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that will be subsequently confirmed plus 1) divided by 30.44. The DR will be calculated for the subgroup of participants with a confirmed objective tumor response.
Progression-Free Survival (PFS) by Independent Expert Review (IER) | Baseline up to progressive disease or death, assessed every 6 weeks (up to 90 weeks)
  PFS is defined as the time in months from start of study treatment to first documentation of objective tumor progression or death due to any cause whichever comes first. PFS is calculated as (first event date minus the date of first dose of study medication plus 1) divided by 30.44. Tumor progression will be determined from radiological image (where data meet the criteria for progressive disease [PD]). IER will be done to re-examine all Investigator assessed outcomes and to provide an independent assessment of response and progression date.
Progression-Free Survival (PFS) by Investigators' Assessment | Baseline up to progressive disease or death, assessed every 6 weeks (up to 90 weeks)
  PFS is defined as the time in months from start of study treatment to first documentation of objective tumor progression or death due to any cause whichever comes first. PFS is calculated as (first event date minus the date of first dose of study medication plus 1) divided by 30.44. Tumor progression will be determined from radiological image (where data meet the criteria for progressive disease [PD]). IER will be done to re-examine all Investigator assessed outcomes and to provide an independent assessment of response and progression date.
Number of Participants With Changes in Tumor Volume | Baseline up to progressive disease or death, assessed every 6 weeks (up to 90 weeks)
  Three dimensional analysis will be used to measure changes in tumor volume.
Number of Participants With Changes in Tumoral Radiological Density | Baseline up to progressive disease or death, assessed every 6 weeks (up to 90 weeks)
  Three dimensional analysis will be used to measure changes in tumoral radiological density.

OTHER OUTCOMES:
Number of Participants With Adverse Events | Baseline up to 30 days after last dose of study drug
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (33):
- United States (21):
  - Sedona, Arizona
  - Denver, Colorado
  - Torrington, Connecticut
  - Indianapolis, Indiana
  - Westminster, Maryland
  - Minneapolis, Minnesota
  - Columbia, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Amsterdam, New York
  - New York, New York
  - Bedford, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Norfolk, Virginia
  - Salem, Virginia
  - Seattle, Washington
  - Spokane, Washington
  - Yakima, Washington
- France (5):
  - Bourdeaux
  - Marseille
  - Saint-Herblain
  - Strasbourg
  - Villejuif
- Israel (4):
  - Jerusalem
  - Rehovot
  - Tel Aviv
  - Tel Litwinsky
- Poland (3):
  - Lubin
  - Rybnik
  - Szczecin

REFERENCES:
- [Derived] Delaloge S, Wolp-Diniz R, Byrski T, Blum JL, Goncalves A, Campone M, Lardelli P, Kahatt C, Nieto A, Cullell-Young M, Lubinski J. Activity of trabectedin in germline BRCA1/2-mutated metastatic breast cancer: results of an international first-in-class phase II study. Ann Oncol. 2014 Jun;25(6):1152-8. doi: 10.1093/annonc/mdu134. Epub 2014 Apr 1. PMID 24692579
- See also: Phase II, Multicenter, Open-label, Clinical Trial of Trabectedin (Yondelis) in Metastatic Breast Cancer Patients With Triple Negative Profile (ER-, PR-, HER2-), HER2 Overexpressing Tumors and BRCA1 or BRCA2 Mutation Carriers — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=779&filename=CR014764_CSR.pdf